CLINICAL TRIAL: NCT01916785
Title: A PROSPECTIVE RANDOMIZED PHASE II STUDY EVALUATING THE OPTIMIZATION OF THE RESIDUAL PLASMATIC LEVEL OF DASATINIB (SPRYCEL®) IN PATIENTS NEWLY DIAGNOSED WITH CHRONIC PHASE CHRONIC MYELOGENOUS LEUKAEMIA (CP-CML).
Brief Title: OPTIM DASATINIB (Optimized Tyrosine Kinase Inhibitors Monotherapy)
Acronym: OPTIM-DASA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Versailles Hospital (Other)
Collaborators: Maisonneuve-Rosemont Hospital (Other); University Hospital, Bordeaux (Other)
Responsible Party: Principal Investigator, Philippe ROUSSELOT, Clinical Coordinator, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2008-006854-17
Record Dates: First submitted 2012-12-18; First posted 2013-08-06 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Myelogenous Leukemia, BCR/ABL Positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A1 (Experimental): Arm A1: Dasatinib dose adjustment based on Cmin ≥3nM value analysed on blood after 7-10 days dasatinib 100mg intake
  Interventions: Drug: Dasatinib
- A2 (Active Comparator): Arm A2: Dasatinib standard dose (100mg/d) with Cmin ≥ 3nM analysed on blood after 7-10 days dasatinib 100mg intake
  Interventions: Drug: Dasatinib
- B (Active Comparator): Arm B : Dasatinib standard dose with Cmin < 3nM analysed on blood after 7-10 days dasatinib 100mg intake
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Dasatinib is a multitargeted tyrosine kinase inhibitor with a 300-fold more potent activity on the BCR-ABL tyrosine kinase in vitro compared to imatinib mesylate
  Other Names: Sprycel®

SUMMARY:
This protocol is a multicentric interventional phase II study from the French CML Intergroup (FILMC).

The core of the protocol is to explore the efficacy and safety of an optimization strategy consisting in the modulation of the dasatinib daily dose according to the results of repeated plasmatic levels of dasatinib.

The objective of this strategy is to improve the overall results of the treatment of early CP-CML in order to avoid the development of resistance and BCR-ABL tyrosine kinase mutations.

The study will be conducted in selected FILMC and Canadian centers.

The study is sponsored by the Hôpitaux de Versailles and supported by Bristol-Myers Squibb. The dasatinib treatment will be provided by Bristol-Myers Squibb until marketing authorization is granted in that indication.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥ 18 years
2. ECOG Performance Status score 0-2
3. Philadelphia chromosome positive newly diagnosed (≤ 3 months) CP-CML
4. patients not previously treated except with hydroxyurea or imatinib (less than 4 weeks for imatinib)
5. Signed written inform consent
6. Adequate hepatic function defined as: total bilirubin ≤ 2.0 times the institutional ULN; ALT and AST ≤ 2.5 times the institutional upper limit of normal (ULN).
7. Adequate renal function defined as serum creatinine ≤ 3 times the institutional ULN.
8. Women of childbearing potential (WOCBP) must be using an adequate method of contraception.

Exclusion Criteria:

1. Patients with BCR-ABL positive, Philadelphia negative CML
2. Patient previously treated with a tyrosine kinase inhibitor (TKI) except with imatinib during less than 4 weeks.
3. Pregnancy
4. Active malignancy
5. Uncontrolled or significant cardiovascular disease
6. Patients with QTc > 450 ms
7. Significant bleeding disorder unrelated to CML
8. Concurrent severe diseases which exclude the administration of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2009-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cumulative rate of significant AE | 12 months therapy
  The cumulative rate of serious AEs defined by grade 3-4 fluid retention, all grade pleural effusion, haematological grade 3-4 AEs related to dasatinib and/or all AE leading to dasatinib discontinuation within the first year of therapy

SECONDARY OUTCOMES:
Rate of treatment interruptions | 12 months therapy
  To compare the rate of treatment interruptions
Cumulative duration of dasatinib interruption | 12 months therapy
  To compare the cumulative duration of dasatinib interruption C. To compare the median dose of dasatinib administered during the first 12 months
Mean dose of dasatinib | 12 months therapy
  To compare the mean dose of dasatinib administered during the first 12 months
Cumulative rate of complete cytogenetic response | 12 months therapy
  To compare the cumulative rate of complete cytogenetic response (CCR) at 6, 12 and 18 months, and every 12 months thereafter
Cumulative rate of major molecular response | 12 months therapy
  To compare the cumulative rate of major molecular response (MMR) at 3, 6, 12, and 18 months, and every 6 months thereafter
Median dose of dasatinib administered | 12 months therapy
  To compare the median dose of dasatinib administered during the first 12 months
Cumulative rate of complete molecular response | 12 months therapy
  To compare the cumulative rate of complete molecular response at 3, 6, 12 and 18 months, and every 6 months thereafter
Time to molecular response | 12 months therapy
  To compare the time to molecular response (major or complete)
Relationship between peak plasmatic level and efficacy | 12 months therapy
  To analyse the relationship between peak plasmatic level (Cmax) and efficacy in the three arms
Relationship between through plasmatic level and efficacy | 12 months therapy
  To analyse the relationship between through plasmatic level (Cmin) and efficacy in the three arms
Progression-free survival at 5 years | 12 months therapy
  To compare the progression-free survival (PFS) at 5 years in the three arms
Overall survival at 5 years | 12 months therapy
  To compare the overall survival at 5 years in the three arms
Lymphocyte populations before and during dasatinib therapy | 12 months therapy
  To analyse lymphocyte populations before and during dasatinib therapy (for French participating centers - see appendix 14).
Rate of sustained major molecular remission after dasatinib discontinuation in patients in complete molecular response | 12 months therapy
  To evaluate the rate of sustained major molecular remission after dasatinib discontinuation in patients in complete molecular response, CMR (undetectable BCR-ABL transcript, BCR-ABL/ABL IS ratio < 1x10-5)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROUSSELOT, Professeur hémato-oncologie, Principal Investigator — Versailles Hospital
Locations (34):
- Canada (10):
  - Southern Alberta Cancer Research Institute, Calgary
  - Hôpital Charles LeMoyne, Greenfield Park
  - Queen elisabeth II Health Sciences Center, Halifax
  - CH Pierre LeGardeur, Lachenaie
  - Moncton City Hospital, Moncton
  - Hôpital Général Juif - Sir. Mortimer B. Davis, Montreal
  - Hôpital Maisonneuve-Rosemont, Montreal
  - Hôpital Royal Victoria, Montreal
  - Hôpital de l'Enfant Jésus - Centre hospitalier affilié universitaire de Québec, Québec
  - Pavillon Hôtel-Dieu de Québec - Centre hospitalier universitaire de Québec, Québec
- France (24):
  - CHU Angers, Angers
  - Hôpital Avicenne, Bobigny
  - Institut Bergonie, Bordeaux
  - Hopital MORVAN, Brest
  - CH René Dubos, Cergy-Pontoise
  - Hôpital d'Instruction de Armées Percy, Clamart
  - Hopital Henri MONDOR, Créteil
  - Hôpital Claude Huriez, Lille
  - CH Lyon Sud, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Hôpital d'Annecy, Metz-Tessy
  - C.H.U. Brabois, Nancy
  - CHU Hoptel dieu, Nantes
  - Hôpital l'Archet 1, Nice
  - CHU Caremeau, Nîmes
  - Hopital Saint Louis, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital St Antoine, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes - Pontchaillou, Rennes
  - Centre René Huguenin, Saint-Cloud
  - Hôpital Purpan, Toulouse
  - CHRU Bretonneau, Tours
  - Central Hospital, Versailles

REFERENCES:
- [Derived] Rousselot P, Mollica L, Guilhot J, Guerci A, Nicolini FE, Etienne G, Legros L, Charbonnier A, Coiteux V, Dartigeas C, Escoffre-Barbe M, Roy L, Cony-Makhoul P, Dubruille V, Gardembas M, Huguet F, Rea D, Cayssials E, Guilhot F, Bergeron A, Molimard M, Mahon FX, Cayuela JM, Busque L, Bouchet S. Dasatinib dose optimisation based on therapeutic drug monitoring reduces pleural effusion rates in chronic myeloid leukaemia patients. Br J Haematol. 2021 Jul;194(2):393-402. doi: 10.1111/bjh.17654. Epub 2021 Jun 30. PMID 34195988